CLINICAL TRIAL: NCT04342962
Title: Tagraxofusp in Patients With CD123+ or With Blastic Plasmacytoid Dendritic Cell Neoplasm Immunophenotype-like Acute Myeloid Leukemia
Brief Title: Tagraxofusp in Patients With CD123+ or With BPDCN-IPh-like Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML2020
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: CD123+ Acute Myeloid Leukemia; Blastic Plasmacytoid Dendritic Cell Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): 12 mcg/kg/day of tagraxofusp for 5 days, for at least 4 cycles of therapy; each cycle is 21 days.
  Patients will receive the study drug until disease progression or in case of toxicity.
  Interventions: Drug: tagraxofusp

INTERVENTIONS:
Drug: tagraxofusp — Tagraxofusp is provided as an intravenous (IV) injectable and administered as a 15-minute IV infusion. Cycle 1 will include a 2-day dosing period for the first 3 enrolled patients (Days 1-2), a 2-day plus an optional 3rd day for patients 4-6 (Days 1-2 + Day 3 if patient meets criteria for continued dosing) and a 3-day dosing period for patients 7 and beyond (Days 1-3). Cycle 2 and beyond will include a 5-day dosing period for all patients (Days 1-5). In all cycles and schedules, dose delays up to Day 10 of each cycle will be allowed for resolution of toxicities.

SUMMARY:
Non-randomized, open-label, multicenter phase II Study for the treatment of

* 25 R/R BPDCN-IF (CD123/CD4/CD56 positive) AML patients and
* 25 patients presenting R/R AML CD123+, but negative for either, or both, CD4 and CD56.

Patients will be treated with 12 mcg/kg/day of tagraxofusp for 5 days, for at least 4 cicles.

ELIGIBILITY:
Inclusion Criteria:

* The patient has evidence of AML in the peripheral blood and/or bone marrow with either BPDCN-IF [CD123/CD4/CD56 (+)] or with AML that is CD123+ but negative for either, or both, CD4 and CD56.
* The patient is ≥18 years old.
* The patient must be refractory to at least one previous line of conventional therapy (either high dose therapy or hypomethylating agents) or relapsed after receiving conventional therapy (a maximum of two previous line of therapy is admitted).
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0 to 2.
* The patient has adequate baseline organ function, including cardiac, renal, and hepatic function:

  1. Left ventricular ejection fraction (LVEF) ≥institutional lower limit of normal as measured by multigated acquisition (MUGA) scan or 2-dimensional (2-D) echocardiography(ECHO) within 21 days before start of therapy and no clinically significant abnormalities on a 12-lead electrocardiogram (ECG).
  2. Serum creatinine ≤1.5 mg/dL (133 μmol/L).
  3. Serum albumin ≥3.2 g/dL (32 g/L) (albumin infusions are not permitted to enable eligibility).
  4. Bilirubin ≤1.5 mg/dL (26 μmol/L).
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal (ULN).
* If the patient is a woman of childbearing potential (WOCBP), she must have a negative serum or urine pregnancy test at screeningwithin 1 week before treatment.
* The patient has signed informed consent before initiation of any study-specific procedures or treatment.
* The patient is able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment.
* The patient (male and female) agrees to use acceptable contraceptive methods for the duration of time on the study and continue to use acceptable contraceptive methods for 1 week after the last infusion of tagraxofusp.

Exclusion Criteria:

* The patient has a diagnosis of acute promyelocytic leukemia (APL; FAB subtype M3).
* The patient has persistent clinically significant toxicities of Grade≥2 from previous chemotherapy (excluding alopecia, nausea, fatigue, and liver function tests [as mandated in the inclusion criteria]).
* The patient has received treatment with chemotherapy, wide-field radiation, or biologic therapy within 14 days of study entry.
* The patient has received treatment with an investigational agent within 14 days of study entry.
* The patient has previously received treatment with tagraxofusp.
* The patient has an active malignancy and/or cancer history (excluding antecedent MDS) that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy will be evaluated on a case by case basis. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease.
* The patient has clinically significant cardiovascular disease (eg, uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months before study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
* The patient has uncontrolled, clinically significant pulmonary disease (eg, chronic obstructive pulmonary disease, pulmonary hypertension) that, in the opinion of the Investigator, would put the patient at significant risk for pulmonary complications during the study.
* The patient has known active or suspected central nervous system (CNS) leukemia. If suspected, CNS leukemia should be ruled out with relevant imaging and/or examination of cerebrospinal fluid.
* The patient is receiving immunosuppressive therapy - with the exception of low-dose prednisone (≤10 mg/day) - for treatment or prophylaxis of graft-versus-host disease (GVHD). If the patient has been on immunosuppressive treatment or prophylaxis for GVHD, the treatment(s) must have been discontinued at least 14 days before study treatment and there must be no evidence of Grade ≥2 GVHD.
* The patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
* The patient is pregnant or breastfeeding.
* The patient has known positive status for human immunodeficiency virus or active or chronic hepatitis B or hepatitis C (Patients with positive serology for HBV can be enrolled and must receive antiviral prophylaxis - i.e lamivudine or entcavir).
* The patient is oxygen-dependent.
* The patient has any medical condition that, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities.
* The patient has AML and requires more than 1 g/day of hydroxyurea (Hydroxyureaispermittedatdoses of ≤1 g/day.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR) | 4 months
  Evaluate the activity of tagraxofusp, in terms of ORR (PR + CR + CRi), in patients with CD123+ or BlasticPlasmacytoid Dendritic Cell Neoplasm-like phenotype (BPDCN-IF) Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML).

SECONDARY OUTCOMES:
Rate of AEs and SAEs | 28 months
  Safety analysis according to CTCAE criteria
Overall survival (OS) | 24 months
  Overall survival
Event Free Survival (EFS) | 24 months
  Event Free Survival
Disease Free Survival (DFS) | 24 months from response assessment
  Disease Free Survival
Cumulative incidence of relapse (CIR) | 24 months from response assessment
  Cumulative incidence of relapse
Percentage of patients undergoing allogeneic stem cell transplantation | 12 months
  in MRD-negative CR

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Aou Policlinico Vittorio Emanuele, Po Ospedaliero "G. Rodolico" - Uo Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Irccs Aou San Martino - Genova - Uo Clinica Ematologica, Genova
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Ad Indirizzo Oncologico, Palermo
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Aou Senese - Uoc Ematologia E Trapianti, Siena